CLINICAL TRIAL: NCT02642848
Title: Clinical Outcomes of Open Wedge High Tibial Osteotomy With Autologous Bone Marrow or Adipose-derived Stem Cell Therapy
Acronym: HTOSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongsik Chae (Other)
Responsible Party: Sponsor-Investigator, Dongsik Chae, Assistant professor, Catholic Kwandong University
Organization: Catholic Kwandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS15OISI0021
Record Dates: First submitted 2015-12-11; First posted 2015-12-30 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis; Genu Varum
MeSH Terms: conditions — Osteoarthritis; Genu Varum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HTO with micro fracture (Active Comparator): High tibial osteotomy(HTO) with micro fracture is an common treatment for the correction of malalignment of the knee treating osteoarthritis.
  Interventions: Procedure: HTO with microfracture
- HTO with bone marrow stem cell (Experimental): High tibial osteotomy(HTO) with transplantation of autologous bone marrow cell concentrate using BMAC collecting from iliac bone.
  Interventions: Procedure: HTO with microfracture; Procedure: Transplantation of bone marrow stem cell
- HTO with adipose derived stem cell (Experimental): High tibial osteotomy(HTO) with autologous adipose-derived stromal vascular fraction transplantation using LipoSculptor collecting from abdominal fat tissue.
  Interventions: Procedure: HTO with microfracture; Procedure: Transplantation of adipose derived stem cell

INTERVENTIONS:
Procedure: HTO with microfracture — High tibial osteotomy(HTO) with micro fracture on femoral condyle is an common treatment for the correction of malalignment of the knee treating osteoarthritis. Device: Tomofix
Procedure: Transplantation of bone marrow stem cell — Transplantation of autologous bone marrow cell concentrate using BMAC collecting from iliac bone. Bone marrow cell cell 6cc
  Arms: HTO with bone marrow stem cell
Procedure: Transplantation of adipose derived stem cell — Transplantation of autologous adipose-derived stromal vascular fraction using LipoSculptor collecting from abdominal fat tissue. Adipose derived stem cell from abdominal fat tissue 3cc
  Arms: HTO with adipose derived stem cell

SUMMARY:
The purpose of this research is to confirm the efficacy of cartilage regeneration (or stem cell transplant) simultaneously performed with high tibial osteotomy. Furthermore, as conventional microfracture surgery on injured cartilage has a disadvantage of the replacement by fibrocartilage, this research intends to prove the excellence over the conventional therapy by proving a hyaline cartilage regeneration of injured cartilage by stem cell.

DETAILED DESCRIPTION:
The prevalence rate of arthritis in medial knee joint is increasing with an increase in senile diseases and there are two main types of therapy: total knee replacement surgery and high tibial osteotomy. Generally, the elderly prefer total knee replacement surgery and younger people prefer high tibial osteotomy. High tibial osteotomy is a procedure to reduce pain and to prevent the progression of osteoarthritis by evenly dispersing excessive load on medial knee joint attributed to varus deformity on the overall knee joint through the correction of abnormal anatomical axis arising from degenerative changes in articular cartilage. The clinical outcomes of high tibial osteotomy are reported as favorable but this high tibial osteotomy has a limitation in terms of the regeneration of injured cartilage. Thus, a research to concurrently perform additional therapy for the regeneration of injured cartilage with the osteotomy was released. Microfracture surgery on injured cartilage, autologous chondrocyte implantation, autologous bone marrow injections and adipose derived stem cell injections are typical examples. However, there is not any solid proof for the excellence of concurrent therapy over a therapy using only the osteotomy in the regeneration of injured cartilage. Therefore, this research is designed to conduct a research to prove the excellence of the direct transplantation of stem cell into injured cartilage over the existing concurrent therapy in the regeneration of injured cartilage. Besides, this research intends to compare the cartilage regeneration capabilities of bone marrow and adipose-derived stem cell.

ELIGIBILITY:
Inclusion Criteria:

15 or more to 65 years of age or younger Classification of degenerative arthritis: Kellgren-Lawrence grade I, III, III Arthritis lesion limited to medial knee joint Varus deformity of knee joint of 15 degrees or less BMI under 35

Exclusion Criteria:

More than 65 years of age Classification of degenerative arthritis: Kellgren-Lawrence grade IV Lesions of arthritis (Kellgren-Lawrence grade III, IV) found in lateral knee joint Varus deformity of knee joint more than 15 degrees BMI above 35 Operation history - Surgery of Microfracture and fracture, and ligament regeneration History of intraarticular injection of steroid and hyaluronic acid in the last 3 months

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Knee score | one year
MRI | One year
  Using MRI, evaluate cartilage conditions by ICRS grade
Arthroscopic finding | One year
  Using arthroscopy, evaluate degree of cartilage repair

CONTACTS AND LOCATIONS:
Locations (1):
- International St. Mary's Hospital, Incheon, Incheon, South Korea